CLINICAL TRIAL: NCT07116837
Title: Perceived Effectiveness of Vaping Prevention Ads Among Adolescents and Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-2140
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaping (Experimental): Adolescents and young adults who are susceptible to vaping or currently vape.
  Interventions: Behavioral: Vaping prevention video ads

INTERVENTIONS:
Behavioral: Vaping prevention video ads — Participants will view and rate 5 vaping prevention video ads. The vaping prevention video ads cover a variety of different topics and were identified in a previous study activity.

SUMMARY:
The purpose of the Aim 2 study is to assess the perceived effectiveness of vaping prevention ads among adolescents and young adults and identify which features of video ads predict perceived message effectiveness. Participants will include adolescents aged 13-17 and young adults aged 18-20 who live in the US and who are susceptible to vaping or who currently vape. In an online survey, participants will be randomized to view five randomly selected vaping prevention ads identified from a previous content analysis. After viewing the videos, participants will rate each video on the perceived message effectiveness scale and respond to questions about vaping appeal and urge to vape. The survey will take 15-20 minutes.

A follow-up survey of a subset of participants will be conducted around two weeks after they have been exposed to vaping prevention video ads in the baseline survey. Participants will view a total of six videos, including the five videos they watched previously, shown one at a time, along with one "decoy" video ad. After watching each video ad, participants will indicate whether they remember seeing the ad in the survey they took around two weeks prior. The survey will take 10-15 minutes.

DETAILED DESCRIPTION:
Health communication campaigns are a scientific approach for preventing and reducing tobacco product use among adolescents. Although a growing number of studies have examined the effects of e-cigarette communication among young adults, there is only a modest number of published studies targeting adolescents. There is little information about the objective features of vaping prevention video ads. Additionally, the follow-up study will explore how ad features are associated with recognition.

Setting: This study is an online survey of adolescents and young adults (age 13-20) who are susceptible to vaping or who currently vape and live in the United States.

Recruitment and Informed Consent: Adolescent and young adult participants will be recruited by Qualtrics Services. Participants who are 18 to 20 years old and are eligible for the study will view a consent form as part of the survey and check a box to indicate that they agree to participate in the study. For minor participants, Qualtrics will recruit parents of 13-17-year-olds, so they will receive the survey invitation with the parental permission/consent form. From there, parents will be asked to pass the survey to their child. Once the participant has completed the consent/assent process, they will be able to begin the survey.

Procedures: up to 3,500 adolescents and young adults who are susceptible to vaping or currently vape will be randomized to view 5 randomly selected ads from a pool of vaping prevention video ads identified from previous study activities. Participants will be screened for susceptibility to vaping or current vape use. Participants will then answer questions on demographic information and tobacco product use. They will view 5 videos, 1 at a time ,randomly assigned from the larger pool of videos. After viewing the videos, participants will rate each video on perceived message effectiveness (primary outcome) and respond to questions about vaping appeal and urge to vape (secondary outcomes). Finally, participants will respond to standard questions on psychological distress, tobacco product use in the home, and general health-related questions. After the survey, participants will view a debrief page with information about tobacco use harms. The survey will take 15-20 minutes.

For the follow-up study, a subset of participants will be asked to complete another survey around two weeks after they have been exposed to vaping prevention video ads in the first survey. In this survey, participants will view a total of six videos, including the five videos they watched when taking the Aim 2 survey around two weeks earlier, shown one at a time, along with one "decoy" video ad. The order of the videos will be randomized. After watching each video ad, participants will indicate whether they remember seeing the ad in the survey they took around two weeks prior. The follow-up survey will take 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-20 years old
* Current vaper (defined as using e-cigarettes in the past 30 days) or susceptible to vaping. Participants will be considered 'susceptible to vaping' if they answer anything other than "definitely not" to 3 screening items assessing their susceptibility to vaping. An example item is, "If one of your best friends were to offer you a vape, would you use it?" (Definitely not, probably not, probably yes, definitely yes).
* Live in the United States

Exclusion Criteria:

• Live outside of the United States

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3500 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Perceived Message Effectiveness | Baseline (Main study)
  The 3-item perceived message effectiveness scale assesses the extent to which participants perceived the vaping prevention video ads as effective. Response options are on a 5-point scale from 1="Not at all" to 5="A great deal". The overall scale score is determined by averaging scores from the 3 items, with higher scores representing higher perceived message effectiveness. This is the primary outcome for the main study.
Recognition | Two-week Follow-up
  This survey item assesses whether the participant remembers viewing the ad in the baseline survey 2 weeks prior. Response options are "Yes", "No", and "Not sure". The response will be dichotomized as 1 = "Yes" and 0 = "No"/"Not sure" for analyses. This is the primary outcome for the follow-up study.

SECONDARY OUTCOMES:
Urge to vape | Baseline
  This survey item assesses the extent to which the video ad makes participants want to vape. Response options are on a 5-point scale from 1="Not at all" to 5="A great deal". A higher score represents a stronger urge to vape. This is a secondary outcome of the main study.
Vaping appeal | Baseline
  This survey item assesses the extent to which the ad makes vaping seem appealing. Response options are on a 5-point scale from 1="Not at all" to 5="A great deal". A higher score represents higher vaping appeal. This is a secondary outcome of the main study.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kowitt, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Seth Noar, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Youjin Jang, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials